CLINICAL TRIAL: NCT04315558
Title: Revefenacin in Acute Respiratory Insufficiency in COPD (RARICO)
Brief Title: Revefenacin in Acute Respiratory Insufficiency in COPD
Acronym: RARICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Theravance Biopharma (Industry); Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Principal Investigator, Igor Barjaktarevic, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#20-000129
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: COPD; Acute Respiratory Failure
Keywords: COPD; Acute Respiratory failure; Long acting muscarinic antagonist; nebulizer; mechanical ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Ipratropium

STUDY DESIGN:
Intervention Model Description: pragmatic, randomized, controlled, double-blinded
Who Masked: Participant, Care Provider, Investigator
Masking Description: blinded medication delivery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Revefenacin (Experimental): Revefenacin will be delivered once daily via nebulizer. In order to allow for full blinding and steady Q6 hours regimen in control arm, at hours 6, 12 and 18 after the Revefenacin dose, nebulized normal saline will be delivered.
  Interventions: Drug: Revefenacin Inhalation Solution [Yupelri]
- Ipratropium (Active Comparator): Nebulized ipratropium will be delivered via nebulizer Q6 hours.
  Interventions: Drug: Ipratropium Bromide

INTERVENTIONS:
Drug: Revefenacin Inhalation Solution [Yupelri] — nebulized drug comparison
  Arms: Revefenacin
Drug: Ipratropium Bromide — nebulized drug comparison
  Arms: Ipratropium

SUMMARY:
RARICO is a pragmatic, randomized, controlled, double-blinded, multi-center trial evaluating the safety and feasibility of nebulized revefenacin in comparison to nebulized ipratropium in patients with COPD and acute respiratory failure requiring invasive mechanical ventilation.

DETAILED DESCRIPTION:
Objective: To assess the efficacy of nebulized revefenacin in improving the lung mechanics of COPD patients with acute respiratory failure requiring invasive mechanical ventilation (MV), in comparison to a control group receiving the short-acting muscarinic antagonist ipratropium.

Hypothesis: Revefenacin is as efficacious as ipratropium in improving the lung mechanics of COPD patients with acute respiratory failure.

Study Design:

RARICO is a pragmatic, randomized, controlled, double-blinded, multi-center trial evaluating the safety and feasibility of nebulized revefenacin in comparison to nebulized ipratropium in patients with COPD and acute respiratory failure requiring invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 40 years of age
* Acute respiratory failure requiring invasive mechanical ventilation
* Documented history of COPD based on spirometric evidence of FEV1/FVC<70%
* Smoking history >10 years (current or prior)
* Invasive mechanical ventilation for < 96 hours

Exclusion Criteria:

* Chronic invasive mechanical ventilation via tracheostomy. Patients with tracheostomy alone without chronic mechanical ventilation may be enrolled.
* Expected duration of mechanical ventilation <24 hours
* Hypersensitivity to muscarinic antagonists
* Inability to tolerate albuterol
* Lack of documented COPD history
* For patients taking short- or long-acting muscarinic antagonists (SAMAs or LAMAs) at the time of screening, inability or unwillingness to undergo the SAMA or LAMA washout period (6 hours or 24 hours, respectively) prior to initiating study drug.
* Presence of ARDS or acute congestive heart failure
* Unwillingness or inability to remain on the study drug with for the duration of the study
* Unwillingness or inability to have open-label muscarinic antagonists withheld for duration of the study
* Unwillingness or inability to utilize the Puritan-Bennett 980 (PB980) ventilator
* Pulmonary comorbidities such as pneumothorax or pneumomediastinum that, in the opinion of the investigator or clinical team, can pose a risk to subject safety or interfere with the subject's ability to complete the study procedures.
* Documented restrictive lung disease or history of interstitial lung disease
* Actual body weight exceeding 1 kg per centimeter of height
* Pregnancy
* AST or ALT > 3 times the upper limit of normal, or other clinically significant acute or chronic liver disease
* Known history of glaucoma
* Enrollment in other interventional clinical trial
* Moribund patient not expected to survive >24 hours
* Decision to withhold life-sustaining treatment, except in those patients committed to full support except cardiopulmonary resuscitation
* Inability to obtain informed consent from patient or legally authorized representative (LAR)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Reduction in total inspiratory resistance Rstat at the time of drug trough | 7 days
  Reduction in total inspiratory resistance across the airways and ventilator circuit measured by the change in Static Resistance (Rstat) at the time of drug trough

SECONDARY OUTCOMES:
Reduction in total inspiratory resistance Rdyn at the time of drug trough | 7 days
  Reduction in total inspiratory resistance across the airways and ventilator circuit measured by the change in Dynamic Resistance (Rdyn) at the time of drug trough
Reduction in Resistive pressure (Pres) at the time of drug trough | 7 days
  Reduction in total inspiratory resistance across the airways and ventilator circuit measured by the change in Resistive pressure (Pres) at the time of drug trough
Reduction in total inspiratory resistance Rstat at the time of drug peak | 7 days
  Reduction in total inspiratory resistance across the airways and ventilator circuit measured by the change in Static Resistance (Rstat) at the time of drug peak
PaCO2 | 7 days
  Arterial partial pressure of CO2 measured at the drug trough
Respiratory therapist time at bedside | 7 days
  RT resource utilization as reflected in the total effective time spent at the bedside providing care
ICU Length of stay | Hospital stay, expected to be less than 28 days
  Time spent in the ICU from the enrollment in the study through the same-stay discharge from the hospital
Ventilator-free days to day 28 | Hospital stay, expected to be less than 28 days
  Time spent ventilator-free from the day of enrollment in the study through the same-stay discharge from the hospital

OTHER OUTCOMES:
Exploratory: Ventilator compliance analysis (ventilator dyssynchrony, pressure-volume curve analysis, expiratory flow curve analysis) | 7 days
  Ventilator compliance analysis (ventilator dyssynchrony, pressure-volume curve analysis, expiratory flow curve analysis)
Safety: Paradoxical bronchospasm, Hypersensitivity reaction, Severe urinary retention not explained by other reasons, Severe constipation not explained by other reasons | 7 days
  Number of episodes of paradoxical bronchospasm, Hypersensitivity reaction, Severe urinary retention not explained by other reasons, Severe constipation not explained by other reasons

CONTACTS AND LOCATIONS:
Overall Officials: Igor Z Barjaktarevic, MD, PhD, Principal Investigator — University of California, Los Angeles; Donald Tashkin, MD, Study Director — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan Medical Center at UCLA, Los Angeles, California
  - Santa Monica UCLA, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donohue JF, Kerwin E, Sethi S, Haumann B, Pendyala S, Dean L, Barnes CN, Moran EJ, Crater G. Revefenacin, a once-daily, lung-selective, long-acting muscarinic antagonist for nebulized therapy: Safety and tolerability results of a 52-week phase 3 trial in moderate to very severe chronic obstructive pulmonary disease. Respir Med. 2019 Jul;153:38-43. doi: 10.1016/j.rmed.2019.05.010. Epub 2019 May 23. PMID 31150963
- [Background] Ferguson GT, Feldman G, Pudi KK, Barnes CN, Moran EJ, Haumann B, Pendyala S, Crater G. Improvements in Lung Function with Nebulized Revefenacin in the Treatment of Patients with Moderate to Very Severe COPD: Results from Two Replicate Phase III Clinical Trials. Chronic Obstr Pulm Dis. 2019 Apr 9;6(2):154-165. doi: 10.15326/jcopdf.6.2.2018.0152. Epub 2019 Apr 9. PMID 30974049
- [Background] Donohue JF, Feldman G, Sethi S, Barnes CN, Pendyala S, Bourdet D, Crater G. Cardiovascular safety of revefenacin, a once-daily, lung-selective, long-acting muscarinic antagonist for nebulized therapy of chronic obstructive pulmonary disease: Evaluation in phase 3 clinical trials. Pulm Pharmacol Ther. 2019 Aug;57:101808. doi: 10.1016/j.pupt.2019.101808. Epub 2019 May 30. PMID 31152911
- [Background] Quinn D, Barnes CN, Yates W, Bourdet DL, Moran EJ, Potgieter P, Nicholls A, Haumann B, Singh D. Pharmacodynamics, pharmacokinetics and safety of revefenacin (TD-4208), a long-acting muscarinic antagonist, in patients with chronic obstructive pulmonary disease (COPD): Results of two randomized, double-blind, phase 2 studies. Pulm Pharmacol Ther. 2018 Feb;48:71-79. doi: 10.1016/j.pupt.2017.10.003. Epub 2017 Oct 4. PMID 28987804
- [Background] Zielinski J. Effects of ipratropium bromide on pulmonary hemodynamics in COPD. Chest. 1995 Oct;108(4):1181-2. doi: 10.1378/chest.108.4.1181-b. No abstract available. PMID 7555146
- [Background] Rezaie N, Shams-Hosseini NS, Kashanizadeh A, Karimi MA. Ipratropium bromide is more effective than Salmeterol - Fluticason combination on O2 saturation patients with COPD. J Res Med Sci. 2013 Aug;18(8):731. No abstract available. PMID 24379853
- [Background] Ogale SS, Lee TA, Au DH, Boudreau DM, Sullivan SD. Cardiovascular events associated with ipratropium bromide in COPD. Chest. 2010 Jan;137(1):13-9. doi: 10.1378/chest.08-2367. Epub 2009 Apr 10. PMID 19363211
- [Background] Khan SY, O'Driscoll BR. Is nebulized saline a placebo in COPD? BMC Pulm Med. 2004 Sep 30;4:9. doi: 10.1186/1471-2466-4-9. PMID 15458566
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Breen D, Churches T, Hawker F, Torzillo PJ. Acute respiratory failure secondary to chronic obstructive pulmonary disease treated in the intensive care unit: a long term follow up study. Thorax. 2002 Jan;57(1):29-33. doi: 10.1136/thorax.57.1.29. PMID 11809986
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Maqsood MH, Rubab K, Maqsood MA. The Role of Revefenacin in Chronic Obstructive Pulmonary Disease. Cureus. 2019 Apr 10;11(4):e4428. doi: 10.7759/cureus.4428. PMID 31245215